CLINICAL TRIAL: NCT02176486
Title: A Phase 1b, Randomized, Double-Blind, Placebo-Controlled, Safety, Tolerability and Pharmacokinetic Study of Multiple Rising Doses of MLN9708 for the Treatment of Subjects With ISN / RPS Class III or IV Lupus Nephritis
Brief Title: Safety, Tolerability and Pharmacokinetics of Multiple Rising Doses of Ixazomib in Lupus Nephritis (LN)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient enrollment, no safety or efficacy concerns
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MLN9708_101; U1111-1152-6999 (Other: WHO); 2014-000125-21 (EudraCT Number); 14/LO/1087 (Registry Identifier: NRES)
Record Dates: First submitted 2014-06-25; First posted 2014-06-27 (Estimated); Results first posted 2019-04-08 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-01

CONDITIONS: Lupus Nephritis
Keywords: Drug Therapy
MeSH Terms: conditions — Lupus Nephritis | interventions — ixazomib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort A: Ixazomib 0.5 milligram (mg) (Experimental): Ixazomib 0.5 mg, capsules, orally, once, on Day 1, 8 and 15 in 28-day cycles, Cycles 1 through 3.
  Interventions: Drug: Ixazomib
- Cohort B: Ixazomib 2 mg (Experimental): Ixazomib 2 mg, capsules, orally, once, on Day 1, 8 and 15 in 28-day cycles, Cycles 1 through 3.
  Interventions: Drug: Ixazomib
- Cohort C: Ixazomib 3 mg (Experimental): Ixazomib 3 mg, capsules, orally, once, on Day 1, 8 and 15 in 28-day cycles, Cycles 1 through 3.
  Interventions: Drug: Ixazomib
- Cohort D: Ixazomib 4 mg (Experimental): Ixazomib 4 mg, capsules, orally, once, on Day 1, 8 and 15 in 28-day cycles, Cycles 1 through 3.
  Interventions: Drug: Ixazomib
- Cohorts A through D: Placebo (Placebo Comparator): Ixazomib placebo-matching capsules, orally, once on Days 1, 8 and 15 in 28-day cycle, Cycles 1 through 3.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ixazomib — Ixazomib capsules.
  Other Names: MLN9708
  Arms: Cohort A: Ixazomib 0.5 milligram (mg); Cohort B: Ixazomib 2 mg; Cohort C: Ixazomib 3 mg; Cohort D: Ixazomib 4 mg
Drug: Placebo — Ixazomib placebo-matching capsules.
  Arms: Cohorts A through D: Placebo

SUMMARY:
The purpose of this study is to characterize the safety and tolerability of ixazomib when administered as multiple oral doses at escalating dose levels in participants with lupus nephritis.

DETAILED DESCRIPTION:
The drug being tested in this study is called ixazomib. Ixazomib is being tested to find a safe and well tolerated dose in participants with lupus nephritis. This study will look at side effects and lab results in participants who take ixazomib, along with the characterization of its pharmacokinetics (PK). This study is designed as a randomized, sequential-panel, multiple rising dose study.

The study will enroll approximately 40 participants. The study population will consist of 4 Cohorts. At least 5 participants (4:1 active:placebo) will be recruited into the 0.5 mg dose group (Cohort A), at least 5 participants (4:1 active:placebo) in the 2.0 mg dose group (Cohort B), 8 participants (6:2 active:placebo) in the 3.0 mg dose group (Cohort C), and 8 participants (6:2 active:placebo) in the 4.0 mg dose group (Cohort D). Participants in each Cohort will be asked to take one capsule on Days 1, 8 and 15 in 28-day cycle, for 3 cycles. PK samples will be collected to measure concentrations of ixazomib. The starting dose in Cohort A will be 0.5 mg followed by administrations of 2, 3 and 4 mg in subsequent cohorts.

This multi-center trial will be conducted in the United States and Europe. The overall time to participate in this study is up to 196 days. Participants will make 19 visits to the clinic during the treatment period and will make follow-up visits monthly for 3 months for follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Is female or male and aged 18 to 75 years, inclusive.
4. Has a diagnosis of systemic lupus erythematosus (SLE) defined by meeting either the 2012 Systemic Lupus International Collaborating Clinics (SLICC) criteria or the American College of Rheumatology (ACR) criteria for the classification of SLE. The 4 criteria required by ACR classification are not required to be present at Screening for eligibility.
5. Has a definite diagnosis of LN based on a kidney biopsy done within 2 year of the Screening Visit which demonstrated International Society of Nephrology/Renal Pathology Society (ISN/RPS) class III, IV or V changes [excluding Class III (C), IV-S (C) and IV-G (C)] or World Health Organization (WHO) 1982 classification Class III,IV or V(excluding Class IIIc and IVd).

   1. If no biopsy was done within 2 year of Screening Visit, biopsy can be done during the screening period as a study procedure.
   2. Co-existence of classes is permitted.
6. Has a renal biopsy demonstrating either ISN/RPS or WHO class V or class V with class 2 nephritis with a UPCR of greater than (>) 3 or the participant has a renal biopsy demonstrating either active ISN/RPS or WHO class III or IV nephritis, defined by either one of the following criteria:

   a) A UPCR* of >=1.0 at Screening OR b) A UPCR* >0.5 at Screening and at least one of the following: i. Active urine sediment in the absence of infection or other cause within 3 months of screening, defined as at least one of the following:
   * >=5 red blood cells (RBC) per high power field, not due to causes other than lupus nephritis.
   * >=5 white blood cells (WBC) per high power field in the absence of infection.
   * Presence of cellular casts. ii. The participant has increased levels (above upper limit of normal [ULN]) serum dsDNA autoantibodies at screening.

   iii. Low complement (either C3 or C4) at Screening (>= 25 percent [%] lower than lower limit of normal [LLN]).

   iv. Biopsy within 3 months prior to screening visit indicating active proliferative lupus glomerulonephritis ISN/RPS class III or IV changes [excluding Class III (C), IV-S (C) and IV-G (C)] or WHO 1982 classification Class III or IV (excluding Class IIIc and IVd), with co-existing Class V permitted.
   * Participants may be re-screened once for urinary sediment, proteinuria or complement levels within 2 weeks of the original screening visit.
   * UPCR value for eligibility will be based on the average UPCR obtained from the 3 specimens collected during screening.
7. Has had an inadequate response, in the judgment of the Investigator, to at least 6 months of an immunosuppressive regimen including single or sequential use of at least one of the following: cyclophosphamide (CYC), mycophenolate mofetil (MMF), mycophenolic acid (MA), or azathioprine (AZA).
8. If the participant is on glucocorticosteroids, must be on stable dose equivalent to 20 mg/day or less of prednisone for at least 2 weeks prior to first dose of study medication. Participant who are on a stable dose equivalent to >20 mg/day and <=30 milligram per day (mg/day) of prednisone may be allowed to the study if reviewed by the adjudication committee and approved by the medical monitor; however, the steroid dose should be tapered.
9. Male participants who are sexually active with women of child bearing potential (WOCBP), even if surgically sterilized (that is, status post-vasectomy), must:

   a) Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug.
10. Female participants who are of child bearing potential must:

    a) Agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent through 90 days after the last dose of study drug.
11. This study permits the re-enrollment of a participant that has discontinued the study as a pre- treatment failure (ie, participant has not been randomized). If re-enrolled, the participant must be re-consented.

    * The re-enrollment of all participants who completed Cohort A and B is permitted to subsequent cohorts (2.0 mg and 3.0 mg dose cohorts) after completion of all cycles including the follow-up period if they had no drug-related adverse events greater than Grade 1, no adverse events greater than Grade 2, continue to meet all inclusion and exclusion criteria, and the Safety Review Committee has reviewed and approved enrollment of the subject into a higher dose cohort.
12. Must be receiving Standard of Care (SOC) treatment with an immunosuppressant drug for the treatment of LN (example, MMF, MA or AZA).

Exclusion Criteria:

1. Has received any investigational compound within 30 days or 5 half-lives, whichever is the longer, prior to Screening or is currently participating in another interventional clinical study.
2. Has received ixazomib, bortezomib, or another proteasome inhibitor in a previous clinical study or as a therapeutic agent.
3. Is a sponsor employee, an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in conduct of this study (example, spouse, parent, child, sibling), or may consent under duress.
4. Has an autoimmune disease other than SLE as their main diagnosis.
5. Has drug-induced SLE.
6. Has severe, active central nervous system (CNS) lupus (British Isles Lupus Assessment Group [BILAG] A or B).
7. Has an estimated eGFR of <30 milliliter per minute per 1.73 m^2 (mL/min/1.73m^2), or is on dialysis, or is expected to have a renal transplant within 1 year of randomization, or has had a renal transplant.
8. Has a severe acute infectious disease (example, untreated active tuberculosis (TB), acute viral hepatitis, human immunodeficiency virus (HIV), untreated latent TB, or infections requiring IV anti-microbial treatment within 2 months preceding the Screening Visit.
9. Has a history of a malignant disease (except successfully treated basal cell carcinoma, squamous cell carcinoma, or cervical carcinoma in situ) within 5 years prior to Screening.
10. Has one of the following laboratory test values:

    1. IgG<75% of LLN
    2. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3 times the central laboratory's ULN
    3. Bilirubin >1.5 x ULN (participants with Gilbert Syndrome with a confirmed diagnosis and documented in the subject's medical record will not be excluded based on this criterion).
    4. Platelets <75,000 per cubic millimeter (/mm^3)
    5. Neutrophils <1500/ mm^3 or > 11,000/ mm^3
    6. Hemoglobin <8 grams per deciliter (g/dL)
    7. Positive for Hepatitis B Surface Antigen.
    8. Positive for Hepatitis C antibody.
11. Has a history of drug or alcohol abuse or dependence (as defined by Diagnostic and Statistical Manual of Mental Disorders, fourth Edition [DSM-IV]) within 1 year prior to the screening visit.
12. If female, the participant is pregnant or lactating or intending to become pregnant before, during, or within 3 months after participating in this study; or intending to donate ova during such time period.
13. If male, the participant intends to donate sperm during the course of this study or for 90 days after the last dose. Male participants planning to father during clinical trial conduct or within 90 days after the last planned dose of trial treatment.
14. Has moderate or severe liver disease (Child-Pugh B or C), and/or positive serological tests for hepatitis B (other than due to prior immunization) or hepatitis C.
15. Is taking excluded medications.
16. Has a history of clinically significant neuropathies of National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v 4.03 Grade 2 or higher.
17. Has been treated with CYC within 4 weeks of the Screening Visit.
18. Has been treated with > 3 g/day of MMF within 4 weeks of the Screening Visit.
19. Has been treated with belimumab, abatacept or tocilizumab within 3 months of the Screening Visit.
20. Has been treated with eprazutumab, alemtuzumab, rituximab or other cell depleting biological agents within 6 months of the Screening Visit.
21. Current symptoms of severe, progressive, or uncontrolled non-SLE related renal, hepatic, hematological, gastrointestinal (including hypomotility and ulcerative/inflammatory conditions), pulmonary, cardiac, neurological, or cerebral disease, or other concomitant medical conditions that, in the opinion of the Investigator, might place the subject at unacceptable risk for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-06-09 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2018-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (35):
- United States (12):
  - La Jolla, California
  - Upland, California
  - Port Charlotte, Florida
  - Evergreen Park, Illinois
  - Brooklyn, New York
  - Great Neck, New York
  - Manhasset, New York
  - New York, New York
  - Middleburg Heights, Ohio
  - Lancaster, Pennsylvania
  - Charleston, South Carolina
  - Jackson, Tennessee
- France (4):
  - Lille, Nord
  - Amiens, Somme
  - Paris
  - Strasbourg
- Germany (7):
  - Frankfurt am Main, Hesse
  - Aachen, North Rhine-Westphalia
  - Düsseldorf, North Rhine-Westphalia
  - Mainz, Rhineland-Palatinate
  - Berlin
  - Essen
  - Freiburg im Breisgau
- Italy (4):
  - Rome, Lazio
  - Turin, Piedmont
  - Pisa, Tuscany
  - Padua, Veneto
- Russia (3):
  - Kazan'
  - Kemerovo
  - Saint Petersburg
- Spain (3):
  - Madrid, Madrid, Communidad Delaware
  - Bilbao, Vizcaya
  - Madrid
- United Kingdom (2):
  - London, London, City of
  - London

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available after applicable marketing approvals and commercial availability have been received, an opportunity for the primary publication of the research has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com/Approach for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 8 investigative sites in the United States, Spain and Russia from 09 June 2014 to 19 January 2018.
Pre-assignment Details: Participants with a historical diagnosis of lupus nephritis (LN) were enrolled to receive ixazomib as multiple rising doses (MRD) of 0.5 milligram (mg) in Cohort A and 2.0 mg in Cohort B. This study was terminated early after the completion of Cohorts A and B due to lack of sufficient enrollment to complete the study.
Groups:
- Pooled Placebo: Ixazomib placebo-matching capsules, orally, once, on Days 1, 8 and 15 in a 28-day cycle from Cycle 1 to Cycle 3.
- Cohort A: Ixazomib 0.5 mg: Ixazomib 0.5 mg, capsules, orally, once, on Days 1, 8 and 15 in a 28-day cycle from Cycle 1 to Cycle 3.
- Cohort B: Ixazomib 2 mg: Ixazomib 2 mg, capsules, orally, once, on Days 1, 8 and 15 in a 28-day cycle from Cycle 1 to Cycle 3.
Period: Overall Study
Arm/Group | Pooled Placebo | Cohort A: Ixazomib 0.5 mg | Cohort B: Ixazomib 2 mg
Started | 3 | 5 | 4
Completed | 3 | 5 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set consisted of all participants who were enrolled and received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pooled Placebo | Cohort A: Ixazomib 0.5 mg | Cohort B: Ixazomib 2 mg | Total
Number analyzed (Participants) | 3 | 5 | 4 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 5 | 4 | 12
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 2 | 8
  Male | 2 | 0 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 4 | 2 | 9
  Unknown or Not Reported | 0 | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 2 | 6
  White | 0 | 1 | 2 | 3
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 4 | 3 | 10
  Spain | 0 | 1 | 0 | 1
  Russia | 0 | 0 | 1 | 1
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 169.3 (0.58) | 167.0 (3.39) | 171.5 (6.56) | 169.1 (4.48)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 88.67 (4.216) | 87.56 (16.891) | 92.43 (7.192) | 89.46 (11.229)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 30.92 (1.441) | 31.40 (5.971) | 31.64 (4.660) | 31.36 (4.399)
Smoking Classification [Count of Participants; unit: Participants]
  Never smoked | 2 | 5 | 2 | 9
  Current smoker | 0 | 0 | 1 | 1
  Ex-smoker | 1 | 0 | 1 | 2
Alcohol Classification [Count of Participants; unit: Participants]
  Never drank | 1 | 4 | 2 | 7
  Current drinker | 2 | 1 | 2 | 5
Consumption of Alcohol [Count of Participants; unit: Participants]
  Drank less than or equal to (<=) 4 drinks per day | 2 | 1 | 2 | 5
  Not reported | 1 | 4 | 2 | 7
Female Reproductive Status [Count of Participants; unit: Participants]
  Surgically sterile | 0 | 2 | 1 | 3
  Female of childbearing potential | 1 | 3 | 1 | 5
  Not applicable (participant were male) | 2 | 0 | 2 | 4
Pharmacogenomics (PGx) Consent Obtained [Count of Participants; unit: Participants]
  PGx was obtained | 3 | 5 | 3 | 11
  PGx was not obtained | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced at Least One Grade Greater Than or Equal to (>=) 2 Treatment Emergent Adverse Event (TEAE)
Time Frame: Baseline up to Day 101 (30 days after last dose of study drug)
Population: The safety analysis set consisted of all participants who were enrolled and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Pooled Placebo | Cohort A: Ixazomib 0.5 mg | Cohort B: Ixazomib 2 mg
Number analyzed (Participants) | 3 | 5 | 4
percentage of participants | 33.3 | 20.0 | 25.0

2. Primary Outcome: Percentage of Participants Who Experienced at Least One Treatment Emergent Serious Adverse Event (SAE)
Time Frame: Baseline up to Day 101 (30 days after last dose of study drug)
Population: The safety analysis set consisted of all participants who were enrolled and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Pooled Placebo | Cohort A: Ixazomib 0.5 mg | Cohort B: Ixazomib 2 mg
Number analyzed (Participants) | 3 | 5 | 4
percentage of participants | 0 | 0 | 0

3. Primary Outcome: Percentage of Participants Who Experienced at Least One AE Leading to Study Drug Discontinuation
Time Frame: Baseline up to Day 168
Population: The safety analysis set consisted of all participants who were enrolled and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Pooled Placebo | Cohort A: Ixazomib 0.5 mg | Cohort B: Ixazomib 2 mg
Number analyzed (Participants) | 3 | 5 | 4
percentage of participants | 0 | 0 | 0

4. Primary Outcome: Percentage of Participants With at Least One Markedly Abnormal Value (MAV) for Hematologic Parameters
Time Frame: Baseline up to Day 168
Population: The safety analysis set consisted of all participants who were enrolled and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Pooled Placebo | Cohort A: Ixazomib 0.5 mg | Cohort B: Ixazomib 2 mg
Number analyzed (Participants) | 3 | 5 | 4
percentage of participants | 0 | 0 | 50.0

5. Secondary Outcome: Change From Baseline in Urine Protein to Creatinine Ratio (UPCR) at Day 84
Time Frame: Baseline and Day 84
Population: The safety analysis set consisted of all participants who were enrolled and received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: milligram per milligram creatinine
Arm/Group | Pooled Placebo | Cohort A: Ixazomib 0.5 mg | Cohort B: Ixazomib 2 mg
Number analyzed (Participants) | 3 | 5 | 4
milligram per milligram creatinine
  Baseline | 1.7567 (1.66796) | 2.6134 (2.11100) | 0.7535 (0.40827)
  Change at Day 84 | -0.1680 (1.03388) | -0.4740 (0.96565) | 0.9943 (0.73183)

6. Secondary Outcome: Change From Baseline in Serum Creatinine (sCR) Level at Day 84
Time Frame: Baseline and Day 84
Population: The safety analysis set consisted of all participants who were enrolled and received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: micromoles per liter (mcmol/L)
Arm/Group | Pooled Placebo | Cohort A: Ixazomib 0.5 mg | Cohort B: Ixazomib 2 mg
Number analyzed (Participants) | 3 | 5 | 4
micromoles per liter (mcmol/L)
  Baseline | 91.347 (18.4019) | 72.488 (54.2779) | 81.770 (31.7708)
  Change at Day 84 | -2.947 (22.2468) | 1.768 (7.3961) | 13.260 (39.2029)

7. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) at Day 84
Time Frame: Baseline and Day 84
Population: The safety analysis set consisted of all participants who were enrolled and received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: milliliter/minute/1.73 square meter
Arm/Group | Pooled Placebo | Cohort A: Ixazomib 0.5 mg | Cohort B: Ixazomib 2 mg
Number analyzed (Participants) | 3 | 5 | 4
milliliter/minute/1.73 square meter
  Baseline | 88.7 (28.11) | 130.0 (62.02) | 103.5 (38.77)
  Change at Day 84 | 6.3 (22.19) | 2.6 (29.26) | -0.5 (19.60)

8. Secondary Outcome: Change From Baseline in Levels of Autoantibodies (Anti-double-stranded Deoxyribonucleic Acid [dsDNA]) at Day 84
Time Frame: Baseline and Day 84
Population: The pharmacodynamics (PD) set consisted of all participants who received study drug and had at least 1 post dose PD measurement. Participants who were evaluable for this measure at given time period for the arm were included in the category.
Measure: Mean (Standard Deviation); unit: international units/milliliter (IU/mL)
Arm/Group | Pooled Placebo | Cohort A: Ixazomib 0.5 mg | Cohort B: Ixazomib 2 mg
Number analyzed (Participants) | 3 | 5 | 4
international units/milliliter (IU/mL)
  Baseline: number analyzed (Participants) | 3 | 4 | 4
  Baseline | 18.7 (12.70) | 34.3 (32.57) | 129.3 (140.66)
  Change at Day 84 | -4.3 (6.03) | 7.5 (9.40) | 9.5 (75.76)

9. Secondary Outcome: Change From Baseline in Complement Protein C3 and C4 at Day 84
Time Frame: Baseline and Day 84
Population: The PD set consisted of all participants who received study drug and had at least 1 post dose PD measurement. Participants who were evaluable for this measure at given time period for the arm were included in the category.
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)
Arm/Group | Pooled Placebo | Cohort A: Ixazomib 0.5 mg | Cohort B: Ixazomib 2 mg
Number analyzed (Participants) | 3 | 5 | 4
milligram per deciliter (mg/dL)
  Complement Protein C3: Baseline | 122.3 (59.47) | 82.2 (23.67) | 110.3 (40.24)
  Complement Protein C3: Change at Day 84 | -20.3 (26.76) | -7.4 (10.50) | -19.5 (13.18)
  Complement Protein C4: Baseline | 29.0 (13.08) | 12.4 (8.26) | 20.0 (9.56)
  Complement Protein C4: Change at Day 84: number analyzed (Participants) | 3 | 5 | 2
  Complement Protein C4: Change at Day 84 | -4.7 (4.73) | -0.8 (1.92) | -6.0 (1.41)

10. Secondary Outcome: Plasma Concentrations of Ixazomib at Each Scheduled Collection Time
Time Frame: Cycle 1 Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose (Cycle length is equal to [=] 28 days)
Population: The pharmacokinetic (PK) set consisted of all participants who received one dose of ixazomib and had at least 1 measurable plasma concentration.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Cohort A: Ixazomib 0.5 mg | Cohort B: Ixazomib 2 mg
Number analyzed (Participants) | 5 | 3
nanogram per milliliter (ng/mL)
  Pre-dose | 0.0000 (0.00000) | 0.0000 (0.00000)
  0.25 hour | 0.0000 (0.00000) | 0.0000 (0.00000)
  0.5 hour | 0.4244 (0.69887) | 2.5033 (4.33590)
  1 hour | 0.6776 (0.68219) | 2.2000 (2.35841)
  1.5 hours | 0.5056 (0.72535) | 2.3400 (2.38627)
  2 hours | 0.5134 (0.52152) | 2.2767 (2.07447)
  4 hours | 0.1082 (0.24194) | 1.1700 (1.01602)
  8 hours | 0.0000 (0.00000) | 0.9967 (0.86327)
  24 hours | 0.0000 (0.00000) | 0.5493 (0.48634)
  168 hours | 0.0000 (0.00000) | 0.0000 (0.00000)

ADVERSE EVENTS:
Time Frame: All AEs that started after the first dose of study drug up to Day 168 (study completion)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Pooled Placebo | Cohort A: Ixazomib 0.5 mg | Cohort B: Ixazomib 2 mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/5 | 1/4
Other Adverse Events (participants affected / at risk) | 3/3 | 5/5 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pooled Placebo (N=3) | Cohort A: Ixazomib 0.5 mg (N=5) | Cohort B: Ixazomib 2 mg (N=4)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) — SAE is not a TEAE since it occurred after 30 days after last dose of study drug.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pooled Placebo (N=3) | Cohort A: Ixazomib 0.5 mg (N=5) | Cohort B: Ixazomib 2 mg (N=4)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Eye inflammation (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyuria (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Systemic lupus erythematosus rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-03-06): https://cdn.clinicaltrials.gov/large-docs/86/NCT02176486/SAP_000.pdf
  • Study Protocol (2017-11-30): https://cdn.clinicaltrials.gov/large-docs/86/NCT02176486/Prot_001.pdf